CLINICAL TRIAL: NCT05229536
Title: A Single-center, Randomized, Double-blind, Parallel Control Phase II Clinical Trial to Evaluate Immunogenicity and Safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in Healthy Volunteers Aged From 3 to 35 Months
Brief Title: Immunogenicity and Safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in Volunteers Aged From 3 to 35 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201719805
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose Group (Experimental): Meningococcal ACYW135 Polysaccharide Conjugate Vaccine, 40μg/dose
  Interventions: Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine
- Low dose Group (Experimental): Received Vaccine: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine, 20μg/dose
  Interventions: Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine — Group 1: 3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 10 µg each of Serogroup A, C, Y, and W135 polysaccharide conjugate.
  Arms: High dose Group
Biological: Meningococcal ACYW135 Polysaccharide Conjugate Vaccine — Group 2: 3/2/1 dose(s) according to age of subjects. Single intramuscular dose contains 5 µg each of Serogroup A, C, Y, and W135 polysaccharide conjugate.
  Arms: Low dose Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine in healthy volunteers aged from 3 months to 35 years.

ELIGIBILITY:
Inclusion Criteria:

* People aged 3-35 months;
* Subject who has not been vaccinated with meningococcal group A and C conjugate vaccine, meningococcal group A polysaccharide vaccine and meningococcal group A and C and haemophilus b conjugate vaccine at the aged of 3-11 months, and who have't given boost immunity above 1 year old, and they all meet the physical examination requirements of the project;
* Infants aged 3-11 months should be full-term (37-42 weeks of gestation) and their birth weight should meet the requirements (2500g ≤ body weight ≤ 4000g);
* The guardian signs the informed consent form;
* The guardian and his family agree to comply with the requirements of the clinical trial protocol;
* Subject who had no history of other live vaccines within 14 days before vaccination and no history of other inactivated vaccines within 7 days;
* Axillary body temperature ≤ 37.0 ℃.

Exclusion Criteria:

* History of severe allergic reactions requiring medical intervention (such as swelling of mouth and throat, dyspnea, hypotension or shock);
* Have a history of allergy to the vaccine or vaccine ingredients (especially those allergic to tetanus toxoid), or have a history of other serious adverse reactions to the vaccine;
* A clearly diagnosed history of thrombocytopenia or other coagulation disorders that may cause contraindications to intramuscular injection;
* Abnormal production process, asphyxia rescue history, or congenital malformation, developmental disorder or serious chronic disease;
* Has serious cardiovascular, liver and kidney diseases or congenital abnormalities and HIV infection;
* Suffer from encephalopathy, uncontrolled epilepsy, convulsion and other progressive nervous system diseases;
* Acute disease, severe chronic disease, acute attack of chronic disease and fever (axillary body temperature ≥ 38.0 ℃) in the past 3 days;
* Plan to participate or be participating in any other drug clinical research;
* The interval between the first dose of test vaccine and meningococcal group A polysaccharide vaccine is less than 28 days;
* According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Immunogenicity study of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine as assessed by positive conversion rate | 30 day after each vaccination
Safety study of Meningococcal ACYW135 Polysaccharide Conjugate Vaccine as assessed by the occurrence of adverse events | 30 day after each vaccination
  Evaluate the incidence of adverse reactions for Meningococcal ACYW135 Polysaccharide Conjugate Vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Rongan Center for Disease Control and Prevention, Liuchow, Guangxi, China

IPD SHARING:
Plan to Share IPD: No